CLINICAL TRIAL: NCT00645957
Title: A Comparison of Redrubber Versus Penrose Drains in the Management of Odontogenic (Dental) Infections
Brief Title: A Comparison of Redrubber Versus Penrose Drains
Acronym: redrubber
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Emory University (Other)
Responsible Party: Principal Investigator, Gary F Bouloux MD, DDS, MDSc, FRACDS, FRACDS, Principal Investigator, Emory University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRB00006249
Record Dates: First submitted 2008-03-05; First posted 2008-03-28 (Estimated); Last update posted 2013-11-21 (Estimated); Status verified 2013-11

CONDITIONS: Odontogenic Infection
Keywords: drainage; irrigation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 2 (Active Comparator): This group will have a red rubber drain(s) placed during surgery. This drain(s) will be irrigated intra and post-operatively
  Interventions: Procedure: red rubber drain
- 1 (Active Comparator): This group will have a penrose drain(s) placed during surgery to facilitate drainage post-operatively. This drain (s) will not be irrigated.
  Interventions: Procedure: penrose drain

INTERVENTIONS:
Procedure: penrose drain — incision and drainage of the infection with placement of a penrose drain
  Arms: 1
Procedure: red rubber drain — incision and drainage of infection and placement of a red rubber drain
  Arms: 2

SUMMARY:
All patients presenting to Grady Memorial Hospital with an odontogenic (dental) infection that requires admission to the hospital and incision and drainage will be eligible for inclusion in this pilot study. The surgical method used for incision and drainage will be determined by the attending surgeon who will operate on the patient. The surgical procedure is a simple and universally standardized involving one or more small incisions in the mouth or in the upper neck and the placement of a drain(s) within the infected area to facilitate continued drainage of pus. Subjects will be randomized to either a red rubber or penrose drain(s). The drains are placed through the mouth or upper neck depending on the location of the infection and typically remain in place until the drainage has stopped (several days). All drains are secured with a single stitch through the gum or skin. The drain(s) will be removed bedside by removing a single suture and gently withdrawing the drain. The timing of this is determined by the clinical picture although this typically occurs within the first week. This is not a painful procedure. Currently some surgeons place red rubber drains which, after placement, allow the infection not only to drain but also be irrigated with saline both during the surgery and in the immediate post-operative period. Other surgeons place penrose drains, which, after placement, continue to allow the infection to drain but cannot be irrigated. Red rubber drains require daily irrigation and as such are labor intensive. Furthermore, drains that are irrigated may continue to drain the saline irrigant in the many hours after irrigation that upon clinical inspection may be difficult to distinguish from sero-sanguinous (pus) drainage. It is daily inspection of the drainage (or lack thereof) which determines the appropriate time to remove the drain(s). This in turn may influence time to discharge and ultimately hospital costs

ELIGIBILITY:
Inclusion Criteria:

* age 16 and older

Exclusion Criteria:

* none

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2008-02; Primary Completion 2011-06 (Actual); Study Completion 2011-06 (Actual)

PRIMARY OUTCOMES:
Resolution of infection | several days

CONTACTS AND LOCATIONS:
Locations (1):
- Grady Memorial Hospital, Atlanta, Georgia, United States